CLINICAL TRIAL: NCT00446095
Title: A Phase I/II Multi-Center, Open Label Trial of the Safety and Efficacy of Fostamatinib in Patients With Relapsed/Refractory B-Cell Lymphoma
Brief Title: Efficacy and Safety Study of Fostamatinib Tablets to Treat B-cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4300C00023; C-935788-009 (Other: Rigel Pharmaceuticals)
Record Dates: First submitted 2007-03-08; First posted 2007-03-12 (Estimated); Results first posted 2014-12-18 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma
Keywords: DLCL; Nodular lymphoma; Mantle cell lymphoma; Syk kinase
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — fostamatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fostamatinib (Experimental)
  Interventions: Drug: fostamatinib

INTERVENTIONS:
Drug: fostamatinib — 200 mg PO BID
  Other Names: R935788, R788, fostamatinib

SUMMARY:
Patients: B-cell lymphoma, refractory, diffuse, nodular, mantle, other Phase I : Two groups of 6 patients, escalating dose tolerability- 28 days Phase II: Three groups of 16 patients (nodular, diffuse large cell, mantle cell plus others). Oral bid dosing with highest tolerable dose until toxicity, progression, or withdrawal

DETAILED DESCRIPTION:
This multicenter, open-label study of fostamatinib will take place in two phases.

Phase I Two cohorts, of 6 patients each, will be sequentially assigned to receive 200 mg (Cohort 1) and 250 mg (Cohort 2) PO bid of R788. Patients will be enrolled at 250 mg bid in Cohort 2 only if < 1/6 patients in Cohort 1 experience dose-limiting toxicity (DLT) during the initial 28-day treatment period. If 2 or more patients in Cohort 1 experience DLT during the initial 28-day treatment period, patients in Cohort 2 will receive 150 mg PO bid.

Patients who do not experience DLT or disease progression may continue treatment at the assigned dose level until disease progression, toxicity or withdrawal. Patients who experience DLT may resume treatment at a lower dose level (dose will be decreased by 50 mg) when the toxicity grade has decreased to ≤ 1. Once all patients in Phase I have completed 28 days of treatment, the optimal dose of fostamatinib, based on safety and anti-tumor activity, will be determined.

Phase II 48 additional patients, 3 groups of 16 patients each, will receive fostamatinib at the optimal biologic dose PO bid until tumor progression, limiting toxicity or withdrawal. Group 1 will consist of patients with diffuse large B-cell lymphoma (DLBCL), Group 2 will consist of patients with follicular lymphoma, and Group 3 will consist of patients with mantle cell lymphoma, mucosa-associated lymphoid tissue (MALT) lymphoma, marginal zone lymphomas, small lymphocytic lymphomas (SLL), and chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be > 18 years old.
2. Patients must be willing and able to give written informed consent by signing an IRB-approved Informed Consent Form prior to admission to this study and must fully understand the requirements of the study and be willing to comply with all study visits and assessments.
3. Patients with relapsed/refractory B-cell malignancy, (DLBCL, follicular lymphoma, mantle cell lymphoma, MALT lymphoma, marginal zone lymphoma, CLL or SLL), who have failed at least one prior treatment regimen and for whom no standard therapy exists; patients who are intolerant of standard therapy or who are not candidates for available standard therapy may also be included.
4. Patients must have measurable disease.
5. Patients may be male or female. Men, if sexually active, must agree to use at least one medically acceptable form of birth control for the duration of the study and for 30 days thereafter. Sexually active women of childbearing potential must have a negative serum pregnancy test, and agree to use two independent methods of birth control for the duration of the study and for 30 days thereafter.

Exclusion Criteria:

1. Patients with T-cell lymphoma or primary CNS lymphoma
2. Patients with a history of malignancy other than lymphoma, except basal cell carcinoma of the skin and in situ cervical carcinoma, if < 2 years since curative treatment
3. Chemotherapy within 4 weeks of Day 1 of treatment (6 weeks for mitomycin C and nitrosoureas)
4. Antibody therapy or lymphoma vaccine therapy within 6 weeks of Day 1
5. Radiotherapy within 2 weeks of Day 1, 4 weeks if to marrow-bearing sites (sternum, pelvis)
6. Any other investigational therapy within 4 weeks of Day 1
7. Significant gastrointestinal disease (Crohn's or ulcerative colitis) or major gastric or small bowel surgery
8. Difficulty swallowing or malabsorption
9. Patients with bone marrow impairment: Hgb < 9.0 g/dL; ANC < 1500/μL; platelets < 75,000/μL
10. Patients with impairment of renal function: creatinine > 2.0 g/dL
11. Patients with abnormal liver function: AST/ALT > 3x ULN (up to 5x ULN with liver involvement); bilirubin > 1.5 mg/dL
12. Patients who have been treated with a CYP3A4 inducer/inhibitor within 1 week prior to Day 1 or who are expected to require treatment with CYP3A4 inducer/inhibitor during the course of the study (Appendix IV)
13. Patients with Karnofsky performance status < 60% (Appendix I)
14. Patients whose life expectancy is < 3 months
15. Patients who are known to be HIV positive
16. Patients who have a history of any other significant medical or physical condition that might impair the patient's well being or preclude full participation in the study
17. Pregnant or nursing females
18. Patients receiving systemic or chronic inhaled steroids, with the exception of intermittent dexamethasone for the treatment of emesis or intermittent steroid inhalers for exacerbations of asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, M.D., Study Director — AstraZeneca
Locations (11):
- United States (11):
  - Research Site, Los Angeles, California
  - Research Site, Stanford, California
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Friedberg JW, Sharman J, Sweetenham J, Johnston PB, Vose JM, Lacasce A, Schaefer-Cutillo J, De Vos S, Sinha R, Leonard JP, Cripe LD, Gregory SA, Sterba MP, Lowe AM, Levy R, Shipp MA. Inhibition of Syk with fostamatinib disodium has significant clinical activity in non-Hodgkin lymphoma and chronic lymphocytic leukemia. Blood. 2010 Apr 1;115(13):2578-85. doi: 10.1182/blood-2009-08-236471. Epub 2009 Nov 17. PMID 19965662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 81 patients with lymphoid malignancy were enrolled from 22 March 2007 until 31 January 2008, of which 13 were in Phase I and 68 in Phase II. This study was conducted by 11 investigators at 11 sites in U.S. Primary efficacy analysis was based on Phase II patients so only results from Phase II are posted.
Pre-assignment Details: There was screening period of up to 21 days, after which if all inclusion/exclusion criteria were met, patients were dosed with fostamatinib treatment for a treatment period of 8 weeks. Patients could then continue treatment until disease progression, toxicity or withdrawal from the study
Groups:
- Phase II: DLBCL: Patients with diffuse large B-cell lymphoma (DLBCL) in Phase II
- Phase II: 250mg R788 BID: Patients who received 250mg R788 orally twice daily (PO BID) in Phase II
- Phase II: Other Lymphomas: Patients with mantle cell lymphoma, mucosa-associated lymphoid tissue (MALT) lymphoma, marginal zone lymphomas, small lymphocytic lymphomas and chronic lymphocytic leukemia (SLL/CLL) in Phase II
- Phase I: 200mg R788 BID: Patients who received 200mg R788 orally twice daily (PO BID) in Phase I
- Phase I: 250mg R788 BID: Patients who received 250mg R788 orally twice daily (PO BID) in Phase I
Period: Phase II (8 Weeks)
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase I: 200mg R788 BID | Phase I: 250mg R788 BID
Started | 23 | 21 | 24 | 0 | 0
Completed | 11 | 18 | 21 | 0 | 0
Not Completed | 12 | 3 | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 9 | 2 | 1 | 0 | 0
Not completed — Ongoing | 0 | 0 | 1 | 0 | 0
Period: Phase I (28 Days)
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase I: 200mg R788 BID | Phase I: 250mg R788 BID
Started | 0 | 0 | 0 | 6 | 7
Completed | 0 | 0 | 0 | 5 | 4
Not Completed | 0 | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase I: 200mg R788 BID | Phase I: 250mg R788 BID | Total
Number analyzed (Participants) | 23 | 21 | 24 | 6 | 7 | 81
Age, Continuous [Mean (Full Range); unit: Years] | 63.0 (63) [41 to 87] | 59.0 (59) [41 to 74] | 62.0 (62) [51 to 77] | 78.5 [70 to 91] | 61 [52 to 80] | 61.5 (61.5) [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 7 | 4 | 5 | 29
  Male | 18 | 13 | 17 | 2 | 2 | 52
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 20 | 19 | 21 | 6 | 5 | 71
  Black/African American | 2 | 0 | 3 | 0 | 1 | 6
  Asian | 0 | 2 | 0 | 0 | 1 | 3
  Other: Russian | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate as Assessed According to the"Revised Response Criteria for Malignant Lymphoma" (Cheson 2007).
Description: Proportion of patients with Complete Response (CR) or Partial Response (PR). Revised Response Criteria for Malignant Lymphoma categorises the response of the treatment of a patient's tumour to; CR: the disappearance of all evidence of disease; PR: ≥ 50% decrease in the sum of the perpendicular diameters (SPD) of the six largest dominant nodes plus no increase in the size of other nodes and no new sites of disease; Stable Disease (SD): less than a PR but not progressive disease; Relapsed Disease or PD: Any new lesion or increase by ≥ 50% of previously involved sites from nadir. Primary efficacy is based on Phase II patients only.
Time Frame: Serial tumor assessments were taken at baseline (within 28 days of the start of treatment), and re-evaluated at Day 57, and every 12 weeks thereafter or to confirm response . (Maximum duration of treatment 511 days, Maximum duration of follow-up 812 Days)
Population: Intention to treat (ITT) population is defined as all patients who received at least one dose of fostamatinib.
Measure: Number; unit: Participants
Groups:
- Phase 1: 200mg and 250mg R788 BID: Patients who received 200mg or 250mg R788 orally twice daily (PO BID) in Phase I
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase 1: 200mg and 250mg R788 BID
Number analyzed (Participants) | 23 | 21 | 24 | 13
Participants | 5 | 2 | 7 | 1

2. Primary Outcome: Clinical Benefit Rate as Assessed According to the "Revised Response Criteria for Malignant Lymphoma" (Cheson 2007).
Description: Proportion of patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD)
Time Frame: Serial tumor assessments were taken at baseline (within 28 days of the start of treatment), and re-evaluated at Day 57, and every 12 weeks thereafter or to confirm response (Maximum duration of treatment 511 days, Maximum duration of follow-up 812 Days)
Population: Intention to treat (ITT) population is defined as all patients who received at least one dose of fostamatinib.
Measure: Number; unit: Participants
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase 1: 200mg and 250mg R788 BID
Number analyzed (Participants) | 23 | 21 | 24 | 13
Participants | 9 | 13 | 14 | 9

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: Time from date of first study drug administration to the date of progressive disease as assessed according to the "Revised Response Criteria for Malignant Lymphoma"(Cheson 2007) or the date of death due to any cause, whichever occurred first.
Time Frame: as for outcome 2
Population: Phase II only as was not collected in Phase I. Intention to treat (ITT) population is defined as all patients who received at least one dose of fostamatinib.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas
Number analyzed (Participants) | 23 | 21 | 24
Days | 83.0 [41.0 to 137.0] | 141.0 [61.0 to 253.0] | 126.0 [64.0 to 169.0]

4. Secondary Outcome: Overall Survival (OS)
Description: OS: Time from date of first study drug administration to the date of death.
Time Frame: Overall survival is measured from the time of first administration of study drug to death. (Maximum duration of treatment 511days, Maximum duration of follow-up 812 Days)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas
Number analyzed (Participants) | 23 | 21 | 24
Days | 166.0 [130.0 to NA] — The upper limit of the 95% CI for the median overall survival was not estimable due to small sample size and too few death events and therefore can't be presented. | NA [NA to NA] — The median overall survival could not be calculated due to too few death events.The upper & lower limits of the 95% CI for the median overall survival were not estimable due to small sample size and too few death events, therefore can't be presented. | NA [NA to NA] — The median overall survival could not be calculated due to too few death events.The upper & lower limits of the 95% CI for the median overall survival were not estimable due to small sample size and too few death events, therefore can't be presented.

ADVERSE EVENTS:
Arm/Group | Phase II: DLBCL | Phase II: 250mg R788 BID | Phase II: Other Lymphomas | Phase I: 200mg R788 BID | Phase I: 250mg R788 BID
Serious Adverse Events (participants affected / at risk) | 14/23 | 7/21 | 10/24 | 6/6 | 3/7
Other Adverse Events (participants affected / at risk) | 22/23 | 21/21 | 24/24 | 6/6 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II: DLBCL (N=23) | Phase II: 250mg R788 BID (N=21) | Phase II: Other Lymphomas (N=24) | Phase I: 200mg R788 BID (N=6) | Phase I: 250mg R788 BID (N=7)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 2 | 1 | 0
Chest Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung Infection Pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumococcal Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea Exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Superior Vena Caval Occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Multifocal motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase II: DLBCL (N=23) | Phase II: 250mg R788 BID (N=21) | Phase II: Other Lymphomas (N=24) | Phase I: 200mg R788 BID (N=6) | Phase I: 250mg R788 BID (N=7)
Anaemia (Blood and lymphatic system disorders) | 5 | 7 | 9 | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 5 | 8 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 7 | 2 | 4 | 1
Tachycardia (Cardiac disorders) | 3 | 0 | 2 | 1 | 1
Conjunctival Haemorrhage (Eye disorders) | 0 | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 10 | 12 | 5 | 5
Nausea (Gastrointestinal disorders) | 5 | 11 | 8 | 0 | 4
Vomiting (Gastrointestinal disorders) | 5 | 4 | 6 | 3 | 3
Constipation (Gastrointestinal disorders) | 4 | 3 | 3 | 1 | 1
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 4 | 4 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 3 | 2 | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 1 | 2
Flatulence (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 13 | 16 | 5 | 3
Pyrexia (General disorders) | 8 | 3 | 7 | 3 | 1
Oedema Peripheral (General disorders) | 4 | 3 | 4 | 5 | 0
Asthenia (General disorders) | 2 | 1 | 1 | 4 | 3
Axillary Pain (General disorders) | 2 | 0 | 1 | 0 | 0
Chills (General disorders) | 2 | 1 | 2 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 5 | 5 | 1 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 1 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 2 | 0 | 2 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 6 | 4 | 3 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 5 | 3 | 0 | 0 | 1
Blood Alkaline Phosphatase Increased (Investigations) | 4 | 3 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 3 | 2 | 0 | 0
Blood Bilirubin Increased (Investigations) | 1 | 1 | 3 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 3 | 0 | 0 | 0
Blood Bicarbonate Increased (Investigations) | 2 | 1 | 0 | 0 | 0
Blood Phosphorus Decreased (Investigations) | 2 | 0 | 2 | 1 | 1
Blood Sodium Decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 2 | 2 | 2 | 0 | 0
Weight Decreased (Investigations) | 2 | 1 | 2 | 4 | 1
White Blood Cell Count Decreased (Investigations) | 1 | 2 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 4 | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Increased Appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 5 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 10 | 8 | 0 | 3
Dizziness (Nervous system disorders) | 1 | 7 | 7 | 3 | 2
Dysgeusia (Nervous system disorders) | 2 | 4 | 2 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 2 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 7 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 9 | 2 | 2
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 2 | 3 | 3 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 1 | 2
Hypertension (Vascular disorders) | 3 | 10 | 7 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 7 | 9 | 11 | 4 | 2
Chest discomfort (General disorders) | 1 | 1 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 2 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 1 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0
Secretion discharge (General disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 3 | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 3 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Multifocal motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Cardioactive drug level increased (Investigations) | 0 | 0 | 0 | 1 | 0
Heart sounds abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 1 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Donor site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This is a small, non-randomized study. Comparisons between the 3 groups cannot be reliably made and should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No